CLINICAL TRIAL: NCT06676839
Title: Effectiveness of the WHO ICOPE (Integrated Care for Older People) Program in Preventing Age-related Functional Decline: a 36-month Randomized Controlled Trial With a 24-month Extension
Brief Title: Effectiveness of the WHO ICOPE (Integrated Care for Older People) Program in Preventing Age-related Functional Decline (ICOPE Trial.Fr)
Acronym: ICOPE Fr
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RC31/23/0597; 2024-A00892-45 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2024-10-15; First posted 2024-11-06 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Ageing
Keywords: ICOPE; PREVENTION; intrinsic capacity; healthy ageing; integrated care; elderly; functional decline; Multi component prevention program

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants, physicians, and healthcare professionals will be informed of the allocation of the subjects' group membership after randomization. However, research nurses who will collect data on the primary and secondary outcomes during visits common to all subjects in the trial will be blinded to the subjects' group assignment. Participants and their caregivers will be asked to avoid mentioning the type of treatment they are receiving to the research nurse conducting the interview.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Participants will receive the complete ICOPE intervention, personalized to their deficit during 60 months (36 months, followed by a 24-month extension)
  The intervention include : 1) a screening (every 6 months), using the ICOPE tool 2) a comprehensive assessment of the 6 functions; 3) a personalized intervention aimed at correcting the trajectory of functional decline, based on the participants' choices and preferences; 4) a follow-up of the intervention. All results are communicated to the primary care physician.
  Follow-up visits take place annually at 12, 24, 36, 48 and 60 months. Data related to the outcomes are collected by the research nurse, blinded to the randomization arm.
  Participants will benefit from telephone follow-up 1.5 months after the inclusion visit and between each visit at 6, 18, 30, 42, and 54 months, to support them in implementing their personalized intervention plan and to collect life events occurred between the 2 visits.
  Interventions: Other: the complete ICOPE program
- Control group (No Intervention): During the comparative phase, participants randomized into the Control group will be referred to their primary care physician to receive usual care tailored to their health status. During the 24 months-extension phase they will benefit from the complete ICOPE as defined in the intervention group.
  Follow-up visits take place annually at 12, 24, 36, 48 and 60 months. Data related to the outcomes are collected by the research nurse, blinded to the randomization arm.
  The team will schedule phone calls for all participants at 6, 18, 30, 42, and 54 months to record life events.
  During the extension phase, participants will benefit from phone call follow-up between each annual visit at 42 months and 54 months, to support their personalized intervention plan.

INTERVENTIONS:
Other: the complete ICOPE program — The participant benefits from a personalized intervention, including 1) a screening to be repeated every 6 months, based on the use of the ICOPE tool, allowing an assessment of the 6 functions necessary for an autonomous lifestyle; 2) a comprehensive assessment step for the 6 functions 3) a personalized intervention step aimed at correcting the trajectory of functional decline, based on the participants' preferences; 4) a follow-up step for this intervention.
  Participants will benefit from telephone follow-up 1.5 months after the start of the program and between each annual visit to support them in implementing their personalized intervention plan.
  At each contact, the ICOPE nurse reviews the participant's implementation of the personalized intervention plan recommendations and their adherence to the program.
  The results of the assessment and the proposed intervention are communicated and discussed with the primary care physician and a summary letter is also sent.
  Arms: Intervention group

SUMMARY:
The World Health Organization (WHO) has designed an integrated care program (ICOPE) aimed at maintaining the functions of elderly people to preserve their autonomy. It includes four steps (Screening, Comprehensive Assessment, Personalized Prevention and Care Plan, Follow-up). The screening tool assesses a person's intrinsic capacity in six key functional domains (mobility, cognition, nutrition, vision, hearing, psychological well-being). This screening can be conducted by a professional or through self-assessment using the digital application (ICOPE Monitor). If a deficit is detected, an alert is issued, and if confirmed by a healthcare professional trained in ICOPE, a comprehensive assessment of the impaired function and a personalized prevention and care plan is proposed by the physician. A trained nurse assists the person in implementing this plan in collaboration with the primary care physician and local professionals. When multiple functions are impaired, it is recommended to conduct a thorough evaluation of all six functions to implement an integrated approach.

The clinical effectiveness of the program in preventing functional decline has not yet been established in a sufficiently long trial.

The investigators propose to evaluate the effect and cost of the ICOPE program in France through a controlled trial. Our hypothesis is that, in the current primary care context, the comprehensive implementation of the program (combining regular screening, comprehensive assessment, prevention and care plan, and follow-up) is necessary to more effectively prevent age-related functional decline compared to the usual care provided by the primary care physician.

DETAILED DESCRIPTION:
ICOPE Trail.Fr is a comparative, multicenter, randomized (1:1), two-arm parallel intervention trial, stratified by center and the number of impairments present at inclusion, open-label, controlled, comparing the effectiveness of the comprehensive ICOPE strategy in preventing functional decline in elderly individuals aged 70 and over living at home, versus the usual care provided by their primary care physician.

Participants will be randomized either 1) into the Intervention group, where they will receive the comprehensive ICOPE intervention program, adapted and personalized to their areas of deficit, or 2) into the Control group, where they will be referred to their primary care physician to receive usual care tailored to their health status.

Follow-up visits take place at the investigator's center at V2 (12 months), V3 (24 months), V4 (36 months), V5 (48 months), and V6 (60 months). Data related to functional scales are collected by the research nurse, who is blinded to the randomization results.

Phone calls will be at 6 (A1), 18 (A2), 30 (A3), 42 (A4), and 54 (A5) months to collect relevant life events.

The intervention duration is 36 months, followed by a 24-month extension phase during which all study participants will receive the comprehensive ICOPE intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 65 years and older.
2. Participants living independently at home (ADL = 6, except for an occasional urinary abnormality which will be accepted).
3. Participants showing functional decline in at least 2 of the 6 functional domains of ICOPE (mobility, cognition, nutrition, vision, hearing, and psychological well-being) identified using the ICOPE screening tool.
4. Participants affiliated with a social protection system.

Exclusion Criteria:

1. Participants who has already benefited from the ICOPE program or who has completed more than one isolated step 1
2. Participants living in a dependent elderly care facility.
3. Participants with a disability preventing them from reaching the trial examination center without assistance (such as dementia or significant mobility impairment).
4. Participants with hearing, visual, or speech impairments preventing them from understanding instructions or communicating with study staff.
5. Participants with a life-threatening illness with a prognosis of less than 5 years.
6. Participants unable to provide informed written consent.
7. Participants under legal protection, guardianship, or trusteeship.
8. Participants participating in another interventional research study.
9. Participants in a relationship with a person participating in the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2031-10-14 (Estimated); Study Completion 2031-10-31 (Estimated)

PRIMARY OUTCOMES:
Functional decline | 36 months
  Global functional decline is a composite measure derived from averaging the Z-score of 6 validated components (mobility : Short Physical Performance Battery), cognition (Mini Mental State Examination), nutrition (Mini Nutritional Assessment), vision (Snellen and Raskin), hearing (Hearing Handicap Inventory for the Elderly-Screening), and psychological well-being (Patient Health Questionnaire-9). Raw scores of each of the 6 tests are converted to Z-scores using means and standard deviations at baseline for each test (to have a same unit for all test).

CONTACTS AND LOCATIONS:
Overall Officials: Laurent BALARDY, MD, Principal Investigator — University Hospital, Toulouse
Locations (6):
- France (6):
  - CHIC, Castres, France
  - Perpignan Hospital, Perpignan, France
  - Bigorre Hospital, Tarbes, France
  - CHU Toulouse, Toulouse, France
  - Angers University hospital, Angers
  - Limoges university hospital, Limoges

IPD SHARING:
Plan to Share IPD: No